CLINICAL TRIAL: NCT02283411
Title: Effectiveness and Safety Study of the Abbott Sensor Based Glucose Monitoring System - Personal and Abbott Sensor Based Glucose Monitoring System - Professional
Brief Title: Effectiveness and Safety Study of the Abbott Sensor Based Glucose Monitoring Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ADC-US-VAL-14135
Record Dates: First submitted 2014-10-31; First posted 2014-11-05 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diabetes Mellitus, Type 1 and Type 2 (Other): Subjects will wear the Abbott Sensor Based Glucose Monitoring Systems and will receive no treatment except for safety purposes.
  Interventions: Device: Abbott Sensor Based Glucose Monitoring System

INTERVENTIONS:
Device: Abbott Sensor Based Glucose Monitoring System — Subjects will wear the Abbott Sensor Based Glucose Monitoring Systems and will receive no treatment except for safety purposes.

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of the Abbott Sensor Based Glucose Monitoring System Personal (System-P) and Abbott Sensor Based Glucose Monitoring System Professional (System-Pro) when used as an adjunct to blood glucose testing over a 14-day wear period in adult subjects. The Abbott Sensor Based Glucose Monitoring System - Professional Sensors will be worn by adult subjects over a 14-day wear period.

The primary objective is to characterize the Systems performance with respect to Yellow Spring Instrument (YSI) reference venous sample measurements. The device performance will be primarily evaluated in terms of point and rate accuracy of the Abbott Sensor Based Glucose Monitoring Systems in reference to YSI.

Safety of the Abbott Sensor Based Glucose Monitoring Systems will be characterized by Adverse Device Effects and Serious Adverse Device Effects experienced by study participants.

240 subjects will be enrolled and additional healthy subjects may also be enrolled in the study as training subjects.

DETAILED DESCRIPTION:
Sensors are inserted into the back of the subject's upper arm for up to fourteen (14) days. The subjects are expected to perform capillary BG tests during the 14-day sensor wear. Three in clinic visits are scheduled during the 14-day sensor wear period. During each in-clinic visit, study staff performed IV blood draws to obtain venous blood for YSI reference glucose measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Subject must have a diagnosis of type 1 or type 2 diabetes mellitus.
3. Use one of the following for their diabetes management:

   * intensive insulin therapy (insulin therapy through an insulin pump and/or multiple daily insulin injections) or
   * non-intensive insulin therapy (Basal insulin, injectable non-insulin anti-diabetic agents such as a pramlintide or GLP-1 agonists, NPH insulin either alone or in combination with regular insulin or fast acting insulin analogue, or oral medication)
4. Intensive-insulin using (IIT) subjects only - During one of the in-clinic sessions, subject is willing to have their blood glucose levels manipulated into high and low glucose levels. Insulin-to-carbohydrate ratio and insulin sensitivity formula must be documented prior to having blood glucose levels manipulated. NIT subjects will only be observed during each in-clinic session.
5. For subjects that exercise routinely (at least 3 times per week), willing to exercise during at least one of the in-clinic sessions, if asked.
6. Willing to perform a minimum of 8 finger sticks per day during the study.
7. Subject must be able to read and understand English.
8. In the investigator's opinion, the subject must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
9. Subject must be available to participate in all study visits.
10. Subject must be willing and able to provide written signed and dated informed consent.

Exclusion Criteria:

1. Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
2. Subject is pregnant, is attempting to conceive or is not willing and able to practice birth control during the study duration (applicable to female subjects only).
3. Subject has extensive skin changes/diseases at the proposed application sites that could interfere with device placement or the accuracy of interstitial glucose measurements. Such conditions include, but are not limited to extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, dermatitis herpetiformis, skin lesions, redness, infection or edema.
4. Subject is on dialysis.
5. Subject has a history of untreated hypothyroidism, adrenal gland failure or insufficiency, celiac disease, renal failure, cystic fibrosis, unstable coronary heart disease, or serious psychiatric disorders.
6. Subjects with a history of hypoglycemia unawareness, hypoglycemic seizures or unconsciousness.
7. Subjects who have experienced diabetes-related complications requiring assistance from another person in the last six months.
8. Subject currently is participating in another clinical trial.
9. Subject has donated blood within 112 days (3.7 months) prior to the beginning of the study activities.
10. Subject is anemic.
11. Subject does not have a known insulin to carbohydrate ratio at the time of enrollment (IIT subjects only).
12. Subject has concomitant medical condition which, in the opinion of the investigator, could interfere with the study or present a risk to the safety or welfare of the subject or study staff. Such conditions include but are not limited to:

    - History of HIV, Hepatitis B or C
13. Subject has X-ray, MRI or CT appointment scheduled during the period of study participation, and the appointment cannot be rescheduled for a time before study participation starts or after study participation ends.
14. Subject has an abnormal EKG, unless cleared for study participation by a cardiologist.
15. Subject is unsuitable for participation due to any other cause as determined by the Investigator.

    Additional Criteria
16. The following subjects may participate in the study but will be excluded from all glycemic and exercise challenges:

    * Subject's taking medications known to mask symptoms or hypoglycemia, such as beta blockers;
    * Subjects with any of the following: clinically significant history of cardiovascular or cerebrovascular disease, cardiac arrhythmia, neurological disorders such as seizures, CVA, or syncope, or hypokalemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Bode, MD, Principal Investigator — Atlanta Diabetes Associates; Ronald Brazg, MD, Principal Investigator — Rainier Clinical Research Center; Kristin Castorino, DO, Principal Investigator — Sansum Diabetes Research Institute; Mark Christiansen, MD, Principal Investigator — Diablo Clinical Research; Douglas Denham, DO, Principal Investigator — Clinical Trials of Texas; David Liljenquist, MD, Principal Investigator — Rocky Mountain Diabetes & Osteoporosis Center
Locations (6):
- United States (6):
  - William Sansum Diabetes Center, Santa Barbara, California
  - Diablo Clinical Research, Walnut Creek, California
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Rocky Mountain Diabetes & Osteoporosis Center, Idaho Falls, Idaho
  - Clinical Trials of Texas, San Antonio, Texas
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Undecided to whether to make individual participant data available.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diabetes Mellitus, Type 1 and Type 2
Started | 156
Completed | 125
Not Completed | 31
Not completed — Withdrawal by Subject | 3
Not completed — Screen Failed | 28

BASELINE CHARACTERISTICS:
Arm/Group | Diabetes Mellitus, Type 1 and Type 2
Number analyzed (Participants) | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 61
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 125

OUTCOME MEASURES:

1. Primary Outcome: The Device Performance Was Evaluated in Terms of Point Accuracy of the Abbott Sensor Based Glucose Monitoring Systems in Reference to Yellow Spring Instrument (YSI).
Description: Point accuracy of the system was evaluated as the proportion of System readings that are within ±20% of the YSI reference value for glucose levels ≥ 80 mg/dL and within ±20 mg/dL for YSI glucose levels <80 mg/dL. All 125 subjects wore both System-P and System-Pro Sensors and were included in the outcome measure. System P, the Personal System which is intended for single patient use and System Pro is intended for use by healthcare professionals (HCP). Each subject had up to 136 YSI samples collected during the study which were paired with sensor glucose readings measured at the same time. Point accuracy of the system was evaluated as the percentage of sensor glucose readings that are within ±20% of the YSI reference value for glucose levels ≥ 80 mg/dL and within ±20 mg/dL for YSI glucose levels <80 mg/dL.
Time Frame: 14 days
Population: A total number of 14284 paired points between sensor glucose readings and YSI glucose are used as the denominator to calculate the percentage of sensor glucose readings that are within ±20% of the YSI reference value for glucose levels ≥ 80 mg/dL and within ±20 mg/dL for YSI glucose levels <80 mg/dL.
Measure: Number; unit: percentage of paired points
Units Other Than Participants: Pairs
Groups:
- Diabetes Mellitus, Type 1 and Type 2: Subjects wore the Abbott Sensor Based Glucose Monitoring Systems (Personal[P] and Professional [Pro] and received no treatment except for safety purposes.
  Abbott Sensor Based Glucose Monitoring System: Subjects wore the Abbott Sensor Based Glucose Monitoring Systems and received no treatment except for safety purposes.
Arm/Group | Diabetes Mellitus, Type 1 and Type 2
Number analyzed (Participants) | 125
Number analyzed (Pairs) | 14284
percentage of paired points
  System Personal | 82.9
  System Professional | 86.4

2. Primary Outcome: Safety of the Abbott Sensor Based Glucose Monitoring Systems Was Characterized by Adverse Device Effects and Serious Adverse Device Effects Experienced by Study Participants.
Description: Safety of the Abbott Sensor Based Glucose Monitoring Systems, including adverse device effects and serious adverse device effects were assessed for all participants enrolled in the study.
Time Frame: Safety was evaluated throughout the subject's study participation.
Population: All 125 subjects who participated in the study are included in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetes Mellitus, Type 1 and Type 2
Number analyzed (Participants) | 125
Participants | 6

3. Secondary Outcome: The Trend Accuracy of the System P Device Performance Was Evaluated.
Description: Trend accuracy of the device performance was assessed by comparing of the glucose rate of change results between the sensor glucose readings and YSI reference results for System P only.
Time Frame: 14 days
Population: A total number of 13566 paired points between sensor glucose readings and YSI glucose are used as the denominator to calculate the absolute difference between the rates of change corresponding to Sensor Reading (GM) and YSI results.
Measure: Number; unit: Percentage of paired points
Units Other Than Participants: Pairs
Arm/Group | Diabetes Mellitus, Type 1 and Type 2
Number analyzed (Participants) | 125
Number analyzed (Pairs) | 13566
Percentage of paired points | 82.8

4. Secondary Outcome: The Temporal System Accuracy at Different Glucose Rates of Change and Different Glucose Ranges (Hypoglycemic, Euglycemic, and Hyperglycemic Ranges) Was Evaluated.
Description: The Continuous Glucose Error Grid Analysis (CG-EGA) in the Hypoglycemic range (YSI ≤ 70 mg/dL), in the Euglycemic range (70 < YSI ≤ 180 mg/dL) and in the Hyperglycemic range (YSI > 180 mg/dL) were evaluated.
Time Frame: 14 days
Population: A total of 13566 paired points between sensor glucose readings and YSI glucose were used to calculate and evaluate the percentage of sensor glucose readings at different glucose rates of change and different glucose ranges (hypoglycemic, euglycemic, and hyperglycemic ranges) in System P only.
Measure: Number; unit: % of paired points
Units Other Than Participants: Pairs
Arm/Group | Diabetes Mellitus, Type 1 and Type 2
Number analyzed (Participants) | 125
Number analyzed (Pairs) | 13566
% of paired points
  in the Hypoglycemic range (YSI ≤ 70 mg/dL) | 86.6
  In the Euglycemic range (70 < YSI ≤ 180 mg/dL) | 97.8
  In the Hyperglycemic range (YSI > 180 mg/dL) | 94.5

5. Secondary Outcome: The Point Accuracy of the Device Performance Was Evaluated in Reference to Capillary Blood Glucose (BG).
Description: Point accuracy of the system was evaluated as the proportion of System readings that are within ±20% of the capillary blood glucose (BG) value for glucose levels ≥ 80 mg/dL and within ±20 mg/dL for capillary blood glucose (BG) levels <80 mg/dL. All 125 subjects wore both System-P and System-Pro Sensors and were included in the outcome measure. System P, the Personal System which is intended for single patient use and System Pro is intended for use by healthcare professionals (HCP). Each subject had approximately112 capillary blood glucose (BG) samples collected during the study which were paired with sensor glucose readings measured at the same time. Point accuracy of the system was evaluated as the percentage of sensor glucose readings that are within ±20% of the BG value for glucose levels ≥ 80 mg/dL and within ±20 mg/dL for BG levels <80 mg/dL.
Time Frame: 14 days
Population: A total number of 11444 paired points between sensor glucose readings and BG glucose are used as the denominator to calculate the percentage of sensor glucose readings that are within ±20% of the BG reference value for glucose levels ≥ 80 mg/dL and within ±20 mg/dL for BG glucose levels <80 mg/dL.
Measure: Number; unit: Percentage of paired points
Units Other Than Participants: Pairs
Arm/Group | Diabetes Mellitus, Type 1 and Type 2
Number analyzed (Participants) | 125
Number analyzed (Pairs) | 11444
Percentage of paired points
  System P | 83.6
  System Pro | 87.8

ADVERSE EVENTS:
Time Frame: up to 45 days
Description: Adverse events assessed for all participants who wore Sensors
Groups:
- Diabetes Mellitus, Type 1 and Type 2: Subjects wore the Abbott Sensor Based Glucose Monitoring Systems (Personal[P] and Professional [Pro] and received no treatment except for safety purposes.
  Reported adverse events were determined to be related to study procedures. Those events were observed in six (6) subjects who wore the two Systems (Personal[P] and Professional [Pro]) as required by protocol.
Arm/Group | Diabetes Mellitus, Type 1 and Type 2
All-Cause Mortality (participants affected / at risk) | 0/125
Serious Adverse Events (participants affected / at risk) | 0/125
Other Adverse Events (participants affected / at risk) | 6/125
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diabetes Mellitus, Type 1 and Type 2 (N=125)
I. V. Blood collection related symptoms (Skin and subcutaneous tissue disorders) | 6 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No